CLINICAL TRIAL: NCT02924077
Title: IMI PROTECT - Work Package 4 - Pregnancy Study: An Exploratory Study of Self-reported Medication Use in Pregnant Women
Brief Title: PROTECT Pregnancy Study: An Exploratory Study of Self-reported Medication Use in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTECT_WP4_v8Mar12
Record Dates: First submitted 2016-09-26; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study was a non-interventional, prospective study of pregnant women who agreed to provide information about their medication use and certain lifestyle factors on a periodic basis throughout their pregnancy. Volunteers were recruited by measures such as placement of pamphlets near pregnancy test kits in pharmacies and by links from carefully selected websites and social networking sites. Subjects were invited to learn about the study either through visiting the study web site or phoning a telephone number where a recorded message described the study and invite eligible women to register for participation.

Participants were asked whether they prefer to provide data via the internet or by interactive voice response system (IVRS).

Data were collected in the predominant natural languages of the four study countries: Denmark, the Netherlands, Poland, and the United Kingdom (UK).

Data were collected on use of prescription and non-prescription medication, as well as on use of herbals and homeopathic medications. More information was be collected from women who provided their response over the internet than by phone, in order to best utilize the full capacity of internet- based data collection.

DETAILED DESCRIPTION:
The PROTECT Pregnancy Study was designed to pilot direct-to-patient data collection methods for use in postmarketing surveillance into the foetal effects of maternal medication use in pregnancy. This study which recruited women between October 2012 and January 2014 explored whether women in participating EU countries were willing to provide information via the internet to enable prospective collection of medication exposure data and information about other life style factors during pregnancy. The study's main objective was to assess the extent to which data collected directly from pregnant women via the Internet and an interactive voice response system (IVRS) would provide information on medication use and other potential risk factors throughout pregnancy that is suitable for research purposes.

Pregnant women were recruited for the study using a variety of methods and were asked about use of medications, alcohol and tobacco, recreational drugs, herbals and other factors that could negatively affect birth outcome. The pilot study revealed that women would indeed volunteer to provide information on medication and lifestyle factors during pregnancy, with 2521 women enrolling from four countries over 8-18 months. The four countries include the United Kingdom (UK), The Netherlands (NL), Denmark (DK) and Poland (PL). Of those who enrolled in the PROTECT pregnancy study, only 2066 provided any data, with all but one providing data via internet.

ELIGIBILITY:
Inclusion Criteria:

* Women who identify themselves as pregnant;
* Access to the internet or telephone for providing data;
* Willingness to provide either their e-mail address or telephone number for automated follow-up reminders;
* Primary residence in one of the four participating EU countries: Denmark, the Netherlands, Poland, and the United Kingdom;
* Proficiency in the predominant natural language of their country of residence : Danish, Dutch, Polish, or English.

Exclusion Criteria:

* Women below the age for providing consent.
* Women who are not resident in one of the four participating countries.
* Women in Denmark who are not willing to provide their civil registration number

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: It was initially planned that a minimum of 1400 pregnant women (5600 women total, study-wide) will be recruited from each of the four participating countries: Denmark, the Netherlands, Poland, and the United Kingdom.
  From this number of 1400 participants per country, a limit of 200 women (800 women total, study-wide) would have contributed data via the phone recording system while 1200 would have participate online.
Sampling Method: Non-Probability Sample
Enrollment: 2521 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy Outcome | At pregnancy end (delivery or termination)
  Patient-reported pregnancy outcome is assessed upon pregnancy termination, stillbirth or live birth, recorded from point of enrollment through 30 days after expected date of confinement. No time to event analyses are performed since the study purpose is to compare self-reported events, including pregnancy outcome, with those same events recorded in electronic medical records and the national pregnancy register in Denmark.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Dreyer, MPH, PhD, Study Director — Quintiles Real-World & Late Phase Reasearch, Cambridge, USA

IPD SHARING:
Plan to Share IPD: No